CLINICAL TRIAL: NCT02085538
Title: A Phase 1, Open-label, Single Dose, Parallel-group Study To Evaluate The Pharmacokinetics Of Palbociclib (Pd-0332991) In Subjects With Impaired Renal Function
Brief Title: Study Of Palbociclib (PD-0332991) In Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A5481014
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Renal Impairment
Keywords: renal impairment; AUC; Cmax; palbociclib; normal matched subjects
MeSH Terms: conditions — Renal Insufficiency | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal Renal Function (Experimental)
  Interventions: Drug: palbociclib
- Mild Renal Impairment (Experimental)
  Interventions: Drug: palbociclib
- Moderate Renal Impairment (Experimental)
  Interventions: Drug: palbociclib
- Severe Renal Impairment (Experimental)
  Interventions: Drug: palbociclib

INTERVENTIONS:
Drug: palbociclib — palbociclib 125 mg oral capsule with food once
  Arms: Normal Renal Function
Drug: palbociclib — palbociclib 125 mg oral capsule with food once
  Arms: Mild Renal Impairment
Drug: palbociclib — palbociclib 125 mg oral capsule with food once
  Arms: Moderate Renal Impairment
Drug: palbociclib — palbociclib 125 mg oral capsule with food once
  Arms: Severe Renal Impairment

SUMMARY:
Since the amount of palbociclib eliminated in urine is 6.9%, renal impairment is not expected to have much impact on palbociclib. However, the Federal Drug Administration (FDA) Guidance recommends a study in subjects with renal impairment when the drug is likely to be used in patients with impaired renal function. Palbociclib is intended for chronic use in cancer patients who may have some degree of impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

* Personally signed and dated informed consent document.
* Renal function calculated by the Cockcroft Gault equation: normal function (CLcr >=90 mL/min), mild: CLcr >=60 mL/min and <90 mL/min, moderate: CLcr >=30 mL/min and <60 mL/min, severe: CLcr <30 mL/min but not requiring hemodialysis.
* Subjects with normal renal function matched for age, weight, gender and race to subjects in impaired renal function groups.

Exclusion Criteria:

* Any condition possibly affecting drug absorption.
* Renal allograft recipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 8 days
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 8 days

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 8 days
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Apparent Oral Clearance (CL/F) | 8 days
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 8 days
Apparent Volume of Distribution (Vz/F) | 8 days
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Plasma Decay Half-Life (t1/2) | 8 days
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Unbound Apparent Oral Clearance (CLu/F) | 8 days
  Clearance of unbound drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the oral bioavailability. Unbound drug clearance is a quantitative measure of the rate at which an unbound drug substance is removed from the blood.
"Unbound Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)u]" | 8 days
  AUC (0 - ∞)u= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞)u for unbound drug. It is obtained from AUC (0 - t)u plus AUC (t - ∞)u for unbound drug.
Unbound Maximum Observed Plasma Concentration (Cmaxu) | 8 days
  Cmaxu is the highest measured unbound plasma concentration during the dosing interval.
"Unbound Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClastu)" | 8 days
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClastu) for unbound drug.
fraction of unbound drug in plasma (fu) | 8 days
  fraction of drug in plasma or tissues that is not bound to plasma or tissue proteins.
Unbound Apparent Volume of Distribution (Vzu/F) | 8 days
  Unbound Volume of distribution is defined as the theoretical volume in which the total unbound amount of drug would need to be uniformly distributed to produce the desired unbound plasma concentration of a drug. Unbound Apparent volume of distribution after oral dose (Vzu/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Avail Clinical Research, LLC, DeLand, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Prism Research, Saint Paul, Minnesota

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481014&StudyName=Study%20Of%20Palbociclib%20%28PD-0332991%29%20In%20Renal%20Impairment